CLINICAL TRIAL: NCT06960811
Title: Study of Association Between Ictal Affective Symptoms, Ictal Consciousness Level and the Presence of Comorbid Epileptic Psychoses
Brief Title: Epileptic Psychoses and Their Link With Ictal Emotions and Consciousness
Acronym: ASPAIC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, TARRADA Alexis, M.D., Central Hospital, Nancy, France
Other Study IDs: 2025PI050-601
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy With Partial Onset Seizures With or Without Secondary Generalization; Psychoses; Epilepsy, Generalized
Keywords: psychoses of epilepsy; postictal psychosis; interictal psychosis; epilepsy; clinical research
MeSH Terms: conditions — Psychotic Disorders; Epilepsy, Generalized; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEP +: Patients diagnosed with epilepsy based on video-EEG recording of seizures and with a psychotic comorbidity according to a standardized psychiatric assessment specialized in Epi-Psy
- PEP -: Patients diagnosed with epilepsy based on video-EEG recording of seizures and without psychotic comorbidity according to a standardized psychiatric assessment specialized in Epi-Psy

SUMMARY:
Background :

Psychiatric comorbidities are common in epilepsy, affecting 50 to 70% of patients, especially when the epilepsy is focal and drug-resistant. Among these comorbidities, psychotic disorders (involving hallucinations and delusions) affect 8% of patients - that is, eight times more frequently than in the general population. Currently, the links between epilepsy and psychotic disorders are poorly understood and often overlooked by physicians, which impacts the mental health care of patients with epilepsy and leads to underdiagnosis.

The aim of this research is to determine whether there are differences in epileptic symptoms between patients with a psychotic comorbidity and those without.

Study design :

The main objective of this research is to better understand whether certain emotional epileptic symptoms are associated with a higher risk of developing psychotic symptoms.

The secondary objectives of this study are to investigate whether the level of consciousness during seizures is associated with a higher risk of developing psychotic symptoms.

To meet these objectives, the study will include patients who (1) have epilepsy, (2) were hospitalized in the video-EEG unit of the Neurology Department at Central Hospital for seizure recording, and (3) underwent a psychiatric evaluation in the context of epilepsy between January 1, 2016, and April 1, 2025.

The study will take place at the University Hospital Center (CHRU) of Nancy, in the Neurology Department, within the video-EEG unit led by Professor Louis Maillard. The research will involve comparing epileptic symptoms between the group of patients without psychosis and the group of patients with psychosis.

Data collection will cover the five days of video-EEG hospitalization, along with information from the psychiatric evaluation, for a total duration of approximately one week per year.

Information for participants:

As part of the routine medical care, data is collected in medical records to ensure appropriate follow-up. For the purposes of this research, data from the medical record will be collected.

No identifying information (such as name, initials, full date of birth, address, or social security number) will be collected.

No additional visits or examinations will be required. Patients will not be contacted or asked to provide any new information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of epilepsy
* Patients hospitalized for at least 5 days for a video-EEG recording
* Patients with a psychiatric evaluation, conducted between 01/01/2016 and 04/01/2025.
* Adult patients able to express their opposition to the use of their data.

Exclusion Criteria:

* Absence of seizure recorded during the video-EEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a certain diagnosis of epilepsy, based on a video-EEG monitoring, hospitalized in tertiary center for epilepsy care, and who have a psychiatric evaluation specialized in patients with epilepsy.
  There are limited exclusion criteria to ensure the best representation of patients with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Ictal emotions | From april 2025 to may 2025
  Clinician-assessment of ictal affective symptomatology (facial, verbal, and motor expression), based on a the visualization of an usual seizure recorded in video-EEG.

SECONDARY OUTCOMES:
Ictal consciousness | From april 2025 to may 2025
  Clinician-rating of the Consciousness Seizure Scale (CSS) validated for the assessment of level of consciousness during a seizure. Scores on the CSS range from 0 to 9, which can be interpreted as follows
  * 0 or 1 meaning a profound alteration of consciousness during seizure
  * 2 to 5 meaning an intermediate alteration of consciousness during seizure
  * 6 and more meaning a relatively preserved consciousness during seizure
Ictal dysautonomy | From april 2025 to may 2025
  Measures of neurovegetatives signs during seizures based on ictal EKG, nurse examination (palor, ...)
Type of aura | From april 2025 to may 2025
  Assessment of the type of aura based on the patients description of their seizure and on the video-EEG recording at the beginning of the seizure

CONTACTS AND LOCATIONS:
Overall Officials: Coraline Hingray, MD, PhD, Study Director — Psychotherapeutic Center of Nancy
Locations (1):
- Center Hospital of Nancy, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarrada A, Aron O, Vignal JP, Ertan D, Maillard L, Hingray C. Anticipatory anxiety of seizures is associated with ictal emotional distress and amygdala onset seizures. Epilepsia. 2022 May;63(5):1130-1140. doi: 10.1111/epi.17215. Epub 2022 Mar 20. PMID 35263805
- [Background] Tarrada A, Hingray C, Sachdev P, Le Thien MA, Kanemoto K, de Toffol B. Epileptic psychoses are underrecognized by French neurologists and psychiatrists. Epilepsy Behav. 2019 Nov;100(Pt A):106528. doi: 10.1016/j.yebeh.2019.106528. Epub 2019 Oct 24. PMID 31654941
- [Background] Hesdorffer DC, Ishihara L, Mynepalli L, Webb DJ, Weil J, Hauser WA. Epilepsy, suicidality, and psychiatric disorders: a bidirectional association. Ann Neurol. 2012 Aug;72(2):184-91. doi: 10.1002/ana.23601. Epub 2012 Aug 7. PMID 22887468